CLINICAL TRIAL: NCT04965077
Title: A Phase I Multicenter, Open Label, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of MIL97 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Treatment of Advanced and Metastatic Solid Tumors With MIL97
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MIL97-CT101
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-12

CONDITIONS: Advanced or Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIL97 (Experimental)
  Interventions: Drug: Recombinant Humanized Monoclonal Antibody MIL97 for Injection

INTERVENTIONS:
Drug: Recombinant Humanized Monoclonal Antibody MIL97 for Injection — Dose escalation phase: The patients confirming to the eligibility criteria will be assigned to the 6 dose groups (0.01mg/kg, 0.03mg/kg, 0.1mg/kg, 0.2mg/kg, 0.3mg/kg 0.45mg/kg, respectively) based on the sequence of inclusion. Each patient will receive an intravenous infusion of MIL97 every 3 week on Day 1 of each cycle. Additional 1 or 2 dose cohorts will receive an intravenous infusion of MIL97 every 2 week on Day 1 of each cycle after last patient finishes DLT observation period.
  Dose expansion phase: One or two recommended expansion doses (either Q3W or Q2W) will be selected from 6 dose groups (0.01mg/kg, 0.03mg/kg, 0.1mg/kg, 0.2mg/kg, 0.3mg/kg 0.45mg/kg) based on results of dose escalation phase. MIL97 will be administered via intravenous infusion for 60 to 90 minutes on Day 1 of each cycle.

SUMMARY:
This is a Phase 1, global, multi-center, open-label, multiple-dose, first-in-human study of MIL97 to evaluate the safety, tolerability, pharmacokinetics, biomarkers and efficacy in subjects with advanced or metastatic solid tumor. The study consists of a dose escalation phase and a dose expansion phase. An accelerated titration design (cohorts 1-2 only) followed by 3+3 dose-escalation design will be used in dose escalation phase.

The starting dose for dose escalation phase is 0.01 mg/kg Q3W, followed by 5 dose cohorts (0.03mg/kg Q3W, 0.1mg/kg Q3W, 0.2mg/kg Q3W, 0.3mg/kg Q3W and 0.45mg/kg Q3W). Duration of dose limiting toxicity (DLT) observation is 21 days. Based on data of 3-week treatment regimen, one or two dose levels may be chosen for Q2w regimen. Duration of dose limiting toxicity (DLT) observation is 28 days.

One or two dose cohorts will be chosen (either 2-week regimen or 3-week regimen cohorts) to expand to total of 10 subjects in each cohort for further exploration of PK as well as safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, >=18 years of age;
2. Diagnosis of Refractory/relapsed metastatic and/or unresectable solid tumors;
3. At least one extracranial measurable unirradiated lesion or evaluable lesion (recist v1.1) ;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1Life expectancy >=3 months;
5. Sufficient organ and bone marrow function within 7 days before enrollment;
6. Life expectancy >=12 weeks;
7. Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion Criteria:

1. have a history of myocardial infarction within 6 months or a history of arterial thromboembolic event within 3 months before the first dose;
2. Comorbidity that would interfere with therapy, including interstitial pneumonia, symptomatic congestive heart failure; unstable angina, uncontrolled hypertension; ongoing cardiac arrhythmia ≥ CTCAE 5.0 Grade 3, active coagulopathy, uncontrolled diabetes, QTcF>450ms (Male) or QTcF>470ms (Female) at screening;
3. Patients have a known or suspected history of an autoimmune disorder, except for the following: Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders such as vitiligo, or alopecia not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are eligible;
4. Have a history of manifested central nervous system (CNS) metastases or have primary brain tumor. Patients with known or suspected leptomeningeal disease or cord compression;
5. Receipt of allograft or allogeneic hematopoietic stem cell transplantation;
6. Patients have another active invasive malignancy, but history of a non-invasive malignancy and history of malignancy that is in complete remission after treatment with curative intent are allowed;
7. Active known clinically serious infections are required intravenous antibiotic treatment;
8. Have a history of primary immunodeficiency, including but not limited with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness;
9. Active and clinical significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C (HCV) (Hepatitis B should be confirmed as HBV surface antigen (HBsAg) positive or HBV core antibody (HBcAb) positive with HBV DNA above ULN);
10. Any antitumor therapy within prior 4 weeks (including chemotherapy, targeted therapy, hormone therapy, immunotherapy, radiotherapy, tumor embolization, etc), except for palliative radiotherapy for relief bone pain;
11. Major surgery within prior 4 weeks or expected to require major surgery during study treatment (Major surgery: laparotomy, thoracotomy, and internal organs excision by laparoscopic surgery);
12. Patients have concurrent received or used an immunosuppressive agent within 14 days before study treatment, with the following exceptions and notes: Systemic steroids at physiologic doses, intranasal, inhaled, topical, intra-articular, and ocular corticosteroids with minimal systemic absorption, transient courses of steroids may be approved by the Medical Monitor;
13. Previous exposure to CD40 antibodies;
14. Patients received a live attenuated vaccine within 28 days before study treatment and plan to receive live vaccines during the study unless approved by both investigator and sponsor;
15. Toxicities due to prior therapy are unresolved to ≤ CTCAE 5.0 Grade 1 except for AEs not constituting a safety risk to the patient based on the judgment of investigators;
16. History of clinically significant sensitivity or allergy to MIL97, their excipients, or intravenous gamma globulin;
17. Females who are pregnant or lactating or who intend to become pregnant during the clinical trial period and within 6 months after discontinuation of study treatment. Female or Male who refused using birth control during the clinical trial period and within 6 months after discontinuation of study treatment;
18. Participation in a therapeutic clinical study within 4 weeks for biological treatments, and within 1 week or 5 half-lives for small-molecule agents, before study drug treatment, or current participation in other therapeutic investigational procedures;
19. Patients who have any clinically significant psychiatric, social, or medical condition that, in the opinion of the investigator, could increase the patient's risk, interfere with protocol adherence, or affect the patient's ability to give informed consent are ineligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of MIL97 treatment-emergent adverse events in patients with advanced or metastatic solid tumor | up to 2.5 year after enrollment
  incidence of AEs and SAEs assessed by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | up to 1.5 year after enrollment
  The area under the curve (AUC) of serum concentration of the drug after the administration
Pharmacokinetics: Cmax; | up to 1.5 year after enrollment
  Maximum concentration (Cmax) of the drug after administration
Objective response rate (ORR); | up to 2.5 year after enrollment
  To evaluate preliminary anti-tumor activity of MIL97 in subjects with advanced or metastatic solid tumor. ORR includes complete remission (CR) and partial remission (PR) assessed by RECIST v1.1 criteria.
Duration of response (DoR); | up to 2.5 year after enrollment
  DOR is defined as the time from the initial response (CR or PR) to the time of disease progression or death, whichever occurs first.
Progression free survival (PFS); | up to 2.5 year after enrollment
  Defined as the time from the first day of study treatment to disease progression or death, whichever occurs first.
The overall survival for patients with advanced or metastatic solid tumor; | up to 2.5 year after enrollment
  Defined as the time from the first day of study treatment to disease progression or death, whichever occurs first.
The Disease control rate for patients with advanced or metastatic solid tumor; | up to 2.5 year after enrollment
  Defined defined as the proportion of patients with objective evidence of CR, PR, or SD.
Immunogenicity; | up to 2.5 year after enrollment
  Anti-Drug Antibodies (ADA) will be tested and percentage of ADA positive patients will be calculated to evaluate immunogenicity of MIL97.
Biomarkers; | up to 2.5 year after enrollment
  measurement of CD80, CD86 and cytokines in human plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China